CLINICAL TRIAL: NCT07002034
Title: A Randomized, Double-Blind, Parallel-Group, Dose-Controlled Study Evaluating the Safety and Efficacy of RE104 for Injection in the Treatment of Adjustment Disorder in Patients With Cancer and Other Medical Illnesses
Brief Title: RE104 Safety and Efficacy Study in Adjustment Disorder in Cancer and Other Medical Illnesses
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reunion Neuroscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RE104-202-ADCO
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Adjustment Disorder
Keywords: Cancer; Amyotrophic Lateral Sclerosis (ALS); Multiple Sclerosis (MS); Parkinson's Disease (PD); Idiopathic Pulmonary Fibrosis (IPF); Depression; Anxiety; Psychiatric Distress
MeSH Terms: conditions — Adjustment Disorders; Neoplasms; Amyotrophic Lateral Sclerosis; Multiple Sclerosis; Idiopathic Pulmonary Fibrosis; Depression; Anxiety Disorders | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1.5 mg RE104 (Active Comparator): A single subcutaneous injection of 1.5 mg RE104 for Injection
  Interventions: Drug: RE104 for Injection
- 30 mg RE104 (Experimental): A single subcutaneous injection of 30 mg RE104 for Injection
  Interventions: Drug: RE104 for Injection

INTERVENTIONS:
Drug: RE104 for Injection — Single, subcutaneous dose of RE104 for Injection

SUMMARY:
The purpose of this study is to determine if treatment with a single dose of RE104 for Injection reduces depressive symptoms or depressive symptoms mixed with anxiety symptoms in participants with Adjustment Disorder due to cancer or other illnesses such as Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), Parkinson's Disease (PD) or Idiopathic Pulmonary Fibrosis (IPF) as compared to active-placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has a ≥4 week history of AjD as defined by DSM-5-TR with either depressed mood, or mixed anxiety and depressed mood confirmed by clinical interview with evidence that the AjD was instigated by one of the following medical illnesses (e.g., diagnosis, impact, management, recurrence, prognosis): Cancer, ALS, MS, PD or IPF
* Is sufficiently ambulatory and capable of self care as necessary to complete study procedures
* Has normal cognitive function
* Is on stable use of antidepressants or psychotherapy, or is willing to delay use until the end of study
* If female is not pregnant or planning to become pregnant. If male is not planning to make a partner pregnant
* Is willing and able to comply with the conditions and requirements of the study

Exclusion Criteria:

* Has a significant risk of suicide
* Has active or medical history of bipolar disorder, schizophrenia, schizoaffective disorder, psychotic disorder and/or borderline personality disorder, or first-degree family history of psychosis or bipolar disorder
* Has active or a history of central nervous system malignancy
* Has other medically significant conditions rendering unsuitability for the study
* Has used or will need to use prohibited medications or therapies
* Has a known sensitivity or intolerance to study intervention or potential rescue medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
RE104 30 mg versus RE104 1.5 mg change from baseline in MADRS total score | Day 7
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity. The total score ranges from 0-60 with higher scores representing greater severity of depression.

SECONDARY OUTCOMES:
RE104 30 mg versus RE104 1.5 mg changes in total score from baseline in Hamilton Anxiety Rating Scale (HAM-A) | Day 7
  The Hamilton Rating Scale for Anxiety (HAM-A) is a 14-item scale that is used to rate the severity of symptoms of anxiety. The total score ranges from 0-56 with higher scores representing greater severity of anxiety.
RE104 30 mg versus RE104 1.5 mg incidence of treatment-emergent adverse events (TEAEs) by frequency, severity and seriousness. | From dosing through study completion (post-dose follow-up is for 42 days)
  A treatment-emergent adverse event (TEAE) is defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pollack, Chief Medical Officer, Study Director — Reunion Neuroscience Inc
Locations (22):
- United States (22):
  - UAB, Psychiatry and Behavioral Neurology, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Kadima Neuropsychiatry Institute, San Diego, California
  - Providence Medical Foundation, Santa Rosa, California
  - University of Colorado, Aurora, Colorado
  - University of South Florida, Department of Psychiatry and Behavioral Neuroscience, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - LSU Health Shreveport, Shreveport, Louisiana
  - Sunstone Therapies, PC, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health, Novi, Michigan
  - University of New Mexico, School of Medicine, Albuquerque, New Mexico
  - NYU Langone Center for Psychedelic Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University, Department of Psychiatry, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Alliance for Multispecialty Research Clinical, Knoxville, Tennessee
  - Dell Medical School, University of Texas at Austin, Austin, Texas
  - Cedar Clinical Research Inc., Draper, Utah
  - UVA Center for Psychiatric Clinical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov